CLINICAL TRIAL: NCT05418426
Title: A Phase 1, Open-Label, Parallel Group Study to Evaluate the Pharmacokinetics and Safety of DARE-HRT1 (80μg Estradiol/4mg Progesterone and 160μg Estradiol/8mg Progesterone Intravaginal Rings) in Healthy PostMenopausal Women
Brief Title: A Phase 1, Open-Label, Parallel Group Study to Evaluate the Pharmacokinetics and Safety of DARE-HRT1 in Healthy PostMenopausal Women
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Daré Bioscience, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: DARE-HRT1-001
Record Dates: First submitted 2022-06-10; First posted 2022-06-14 (Actual); Results first posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2023-08

CONDITIONS: Vulvovaginal Atrophy; Vasomotor Symptoms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- IVR: estradiol 80 ug/day + progesterone 4mg/day (Experimental): 28-day IVR 80/4
  Interventions: Device: IVR Dose 1
- IVR: estradiol 160 ug/day + progesterone 8mg /day (Experimental): 28-day IVR 160/8
  Interventions: Device: IVR Dose 2
- Oracle Estrace(R)/Prometrium(R) (Active Comparator): 29 days (estradiol 1mg/progesterone 100 mg oral capsule)
  Interventions: Drug: Oral Reference

INTERVENTIONS:
Device: IVR Dose 1 — Estradiol 80 ug/progesterone 4 mg
  Arms: IVR: estradiol 80 ug/day + progesterone 4mg/day
Device: IVR Dose 2 — Estradiol 160ug/progesterone 8 mg
  Arms: IVR: estradiol 160 ug/day + progesterone 8mg /day
Drug: Oral Reference — estradiol 1mg/progesterone 100 mg
  Arms: Oracle Estrace(R)/Prometrium(R)

SUMMARY:
An open-label study to assess the PK of estradiol, estrone and progesterone from the DARE-HRT1 intravaginal rings at two different dose strengths.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women with body mass index >/= 18 and </= 38 kg/m2
* Normal cervix and vagina
* An intact uterus
* An acceptable results from an endometrial biopsy
* normal mammogram report within 24 months of screening

Exclusion Criteria:

Prior abnormal cervical screening test (CST) or Pap result within 2 years of screening. Subject can have atypical squamous cells of undetermined significance (ASCUS), if HPV negative.

Subjects with any self-reported active sexually transmitted disease and/or evidence of infection based on visual vaginal exam by the investigator

Subjects with a UTI during screening as assessed by urine dipstick test with abnormal test findings (any positive result for leukocytes AND any positive result for nitrites)

Subjects with > 4 mm endometrium lining at screening (on the transvaginal ultrasound)

Have a history of endometrial hyperplasia or cervical or uterine carcinoma

Subjects with indwelling catheters or requiring intermittent catheterization

Subjects with multiple or unsuccessful (e.g., still having symptoms) pelvic reconstructive surgery, or suffers from pelvic relaxation

Subjects who have had a hysterectomy

Subjects taking any estrogen and/or progesterone products (see Section 4.1 for washout requirements)

Subjects with concomitant use of personal lubricants (water-based lubricants are allowed) or any intravaginal product or medication, either by prescription or over-the-counter (e.g., Femring [estradiol acetate vaginal ring], ESTRING® [estradiol vaginal ring]) with the exception of those who agree not to use these products during the IVR use period

Self-reported or observed vaginal irritation; vaginal, vulvar, or cervical lesions, undiagnosed vaginal bleeding; or tenderness

Subjects with a finding of clinically significant uterine fibroids at screening

Subjects with a known hypersensitivity to progesterone, estradiol, Femring, or the components of the IVR (e.g., ethylene vinyl acetate)

Subjects with known hypersensitivity to peanuts (Prometrium capsules contain peanut oil)

Subjects with prior pelvic malignancies

Subjects with a history of any severe acute or chronic medical or psychiatric condition or laboratory abnormality that could increase the risk associated with trial participation or study treatment administration or could interfere with the interpretation of trial results and, in the judgment of the investigator, would make the subject inappropriate for entry into the trial. This includes but is not limited to the following:

Human immunodeficiency virus (HIV) infection (confirmed by medical history/ serology testing)

Active chronic hepatitis B or hepatitis C infection including hepatitis B surface antigen and hepatitis C antigen positive subjects with or without abnormal liver enzymes (confirmed by medical history/serology testing)

Concurrent neurodegenerative disease

Cardiovascular: uncontrolled hypertension, unstable angina, myocardial infarction or symptomatic congestive heart failure within the past 6 months, serious uncontrolled cardiac arrhythmia, use of Class 1 antiarrhythmic medications, or history of venous thromboembolism or stroke

Dementia or significantly altered mental status that would prohibit the understanding or rendering of informed consent and compliance with the requirements of the protocol

History of gallbladder disease unless gallbladder removed

Symptomatic bacterial vaginosis

Have fasting triglyceride of > 300 mg/dL and/or total cholesterol of > 300 mg/dL

AST or ALT > 1.5 times the upper limit of normal

Fasting glucose > 125 mg/dL

Evidence of current alcohol or drug abuse in the past 60 days including a positive result from the urine drugs of abuse or alcohol screen, or history of drug or alcohol dependence in the last two years, as assessed by principal investigator. Alcohol abuse is defined as greater than 14 standard units/week for females and drug abuse is defined as known psychiatric or substance abuse disorder that would interfere with participation with the requirements of this study, including current use of any illicit drugs.

Participation in any other investigational drug or device trial in which administration of an investigational study drug/device occurred within 30 days or placement of a non-drug eluting medical device within 15 days prior to screening.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Must be female.
Enrollment: 34 (Actual)
Dates: Start 2020-08-18 (Actual); Primary Completion 2021-04-27 (Actual); Study Completion 2022-01-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Friend, PhD, Study Director — Dare Bioscience
Locations (2):
- Australia (2):
  - PARC Clinical Research, Melbourne
  - Keogh Institute for medical Research, Nedlands

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | IVR: Estradiol 80 ug/Day + Progesterone 4mg/Day | IVR: Estradiol 160 ug/Day + Progesterone 8mg /Day | Oracle Estrace(R)/Prometrium(R)
Started | 10 | 12 | 12 (One participant was randomized but was terminated prior to first dose due to protocol violation.)
Completed | 10 | 10 | 11
Not Completed | 0 | 2 | 1
Not completed — Adverse Event | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0
Not completed — Protocol Violation | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | IVR: Estradiol 80 ug/Day + Progesterone 4mg/Day | IVR: Estradiol 160 ug/Day + Progesterone 8mg /Day | Oracle Estrace(R)/Prometrium(R) | Total
Number analyzed (Participants) | 10 | 12 | 11 | 33
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 8 | 12 | 11 | 31
  >=65 years | 2 | 0 | 0 | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.8 (6.66) | 56.0 (3.72) | 57.2 (4.42) | 57.2 (4.97)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 12 | 11 | 33
  Male | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 10 | 12 | 11 | 33
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 10 | 11 | 11 | 32
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  Australia | 10 | 12 | 11 | 33
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 28.2 (3.20) | 29.3 (4.98) | 28.2 (3.18) | 28.6 (3.86)

OUTCOME MEASURES:

1. Primary Outcome: To Determine the Steady State Concentration (Css) for Estradiol
Description: To describe the Pharmacokinetic parameters of estradiol in dose combinations (Estradiol 80 ug/progesterone 4/mg day and Estradiol 160 ug/progesterone 8/mg day)
Time Frame: 28 days
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg/mL
Arm/Group | IVR: Estradiol 80 ug/Day + Progesterone 4mg/Day | IVR: Estradiol 160 ug/Day + Progesterone 8mg /Day | Oracle Estrace(R)/Prometrium(R)
Number analyzed (Participants) | 10 | 12 | 11
pg/mL | 14.4 (83.8) | 29.7 (28.23) | 33.8 (31.5)

2. Primary Outcome: To Determine the Stead State Concentration (Css) for Estrone
Description: To describe the Pharmacokinetic parameters of estrone in dose combinations (Estradiol 80 ug/progesterone 4/mg day and Estradiol 160 ug/progesterone 8/mg day)
Time Frame: 28 days
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg/mL
Arm/Group | IVR: Estradiol 80 ug/Day + Progesterone 4mg/Day | IVR: Estradiol 160 ug/Day + Progesterone 8mg /Day | Oracle Estrace(R)/Prometrium(R)
Number analyzed (Participants) | 10 | 12 | 11
pg/mL | 21.6 (75.0) | 20.4 (48.7) | 199 (32.4)

3. Primary Outcome: To Determine the Steady State Concentration (Css) for Progesterone
Description: To describe the Pharmacokinetic parameters of progesterone in dose combinations (Estradiol 80 ug/progesterone 4/mg day and Estradiol 160 ug/progesterone 8/mg day)
Time Frame: 28 days
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg/mL
Arm/Group | IVR: Estradiol 80 ug/Day + Progesterone 4mg/Day | IVR: Estradiol 160 ug/Day + Progesterone 8mg /Day | Oracle Estrace(R)/Prometrium(R)
Number analyzed (Participants) | 10 | 12 | 11
pg/mL | 1.31 (14.72) | 2.03 (23.90) | 0.501 (90.8)

ADVERSE EVENTS:
Time Frame: Adverse Events were collected from time of signing informed consent until last study visit, approximately 2 months.
Arm/Group | IVR: Estradiol 80 ug/Day + Progesterone 4mg/Day | IVR: Estradiol 160 ug/Day + Progesterone 8mg /Day | Oracle Estrace(R)/Prometrium(R)
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 8/10 | 9/12 | 8/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IVR: Estradiol 80 ug/Day + Progesterone 4mg/Day (N=10) | IVR: Estradiol 160 ug/Day + Progesterone 8mg /Day (N=12) | Oracle Estrace(R)/Prometrium(R) (N=12)
Ear Pain (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Dry Eye (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 2 (2) | 2 (4) | 1 (1) — Inclusive of Upper and Lower abdominal pain
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Discomfort (General disorders) | 0 (0) | 1 (12) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 1 (1)
Injection Site Discomfort (General disorders) | 1 (1) | 0 (0) | 1 (1)
Allergy to arthropod sting (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Tinea pedis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Viral Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Vulvovaginal candidiasis (Infections and infestations) | 2 (2) | 1 (1) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Headache (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 2 (3)
Sensory disturbance (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Euphoric mood (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Breast pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Breast tenderness (Reproductive system and breast disorders) | 1 (1) | 2 (3) | 0 (0)
Dysmenorrhea (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Dyspareunia (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Intermenstrual bleeding (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Nipple pain (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Pelvic discomfort & pain (Reproductive system and breast disorders) | 2 (2) | 3 (3) | 2 (2)
Sexual dysfunction (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Vaginal discharge (Reproductive system and breast disorders) | 2 (2) | 1 (1) | 1 (1)
Vaginal hemorrhage (Reproductive system and breast disorders) | 2 (2) | 3 (3) | 1 (1)
Vulvovaginal burning sensation (Reproductive system and breast disorders) | 2 (2) | 3 (4) | 0 (0)
Vulvovaginal dryness (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Vulvovaginal pain (Reproductive system and breast disorders) | 1 (1) | 1 (3) | 0 (0)
Vulvovaginal pruritus (Reproductive system and breast disorders) | 2 (2) | 2 (3) | 0 (0)
Vulvovaginal swelling (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Hemorrhage (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Hot flush (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
One participant randomized into the Oral Reference group was never dosed as the participant was terminated due to a protocol violation.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI unable to publish trial results after the trial is completed without prior approval from Sponsor.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-03-06): https://cdn.clinicaltrials.gov/large-docs/26/NCT05418426/Prot_SAP_000.pdf